CLINICAL TRIAL: NCT06358534
Title: The Effect of Acceptance and Commitment Therapy-based Psychoeducation Given to Chronic Renal Failure Patients on Illness Adaptation, Psychological Resilience and Life Satisfaction
Brief Title: The Effect of Acceptance and Commitment Therapy in Patients With Chronic Renal Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Kubra Berber, LECTURER, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTEU-SBF-KB-01
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Acceptance and Commitment Therapy; Psychiatric Nursing; psychological flexibility
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: pretest-posttest, control and intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control groups (No Intervention): No intervention was performed in chronic renal failure patients with eGFH values below 29 ml/dl/1.72m.
- intervention groups (Experimental): An 8-session acceptance and commitment therapy-based psychoeducation was applied to chronic renal failure patients with eGFH values below 29 ml/dl/1.72m
  Interventions: Behavioral: psychoeducation based on acceptance and commitment therapy

INTERVENTIONS:
Behavioral: psychoeducation based on acceptance and commitment therapy — psychoeducation based on acceptance and commitment therapy prepared by the researchers was applied individually to the patients
  Arms: intervention groups

SUMMARY:
Psychological flexibility, life satisfaction and adaptation to the disease of individuals with chronic kidney disease were increased with psychoeducation based on acceptance and commitment therapy to be given to individuals with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic renal failure is a condition that affects the kidneys and has long-term consequences for physical, psychological, and social well-being. It reduces quality of life, productivity, and independence, leading to increased costs and the need for care. In order to ensure treatment compliance and maintain living standards, it is important to enhance individuals' readiness for treatment. While there are psychological intervention studies during the treatment process, there are few studies that focus on psychological readiness before dialysis. This study highlights acceptance and determination-based approaches to help individuals become aware of their feelings and thoughts and accept them, minimizing resistance to treatment and improving treatment compliance. By managing negative emotions and thoughts towards the treatment, this study aims to increase disease compliance, provide psychological support during pre-dialysis trainings, diversify the use of acceptance and commitment therapy-based approaches, and promote psychosocial support in chronic diseases in psychiatric nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate in the research
* Diagnosis of CKD Stage 4-5
* GFR below 29ml/min/1.72m2
* 18 years of age and over
* Being literate
* No barriers to verbal communication
* No psychiatric treatment

Exclusion Criteria:

* Receiving haemodialysis and peritoneal dialysis treatment,
* Pregnancy
* The presence of a psychiatric disorder requiring treatment,
* Individuals with transplantation and rejection transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Disease Adaptation Scale (CHAS): | 8 weeks
  The scale, which consists of three sub-dimensions (physical adaptation, social adaptation, psychological adaptation) and 25 items, is a 5-point Likert scale (1: Strongly Disagree, 2: Disagree, 3: Undecided, 4: Agree, 5: Strongly Agree).The total score obtained from the scale is 125. The increase in the scores obtained from the sub-dimensions and/or the whole scale means that the patients' level of adaptation to the disease increases.
Acceptance and Action Questionnaire-II Scale (AAQ-II) | 8 weeks
  The KEF-II is a 7-point Likert-type self-report scale consisting of a total of 7 items. Scale items are graded from 1 ("Never true") to 7 ("Always true"). The lowest score that can be obtained from the scale is 7 and the highest score is 49. Higher total scores indicate an increase in the level of psychological rigidity, while lower scores indicate an increase in the level of psychological flexibility.
Life Satisfaction Scale | 8 weeks
  The scale consisting of five questions is in the form of a five-point Likert scale ranging from '1=not at all appropriate' to '5=very appropriate'. The lowest score that can be obtained from the scale, which has no sub-dimensions, is 5 and the highest score is 25. The high score obtained from the scale indicates a high degree of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: kübra berber, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Health Sciences, Rize, Güneysu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No